CLINICAL TRIAL: NCT05785117
Title: Effect of Non-invasive Auricular Vagal Nerve Stimulation Versus Circuit Weight Training on Nutritional Modulation in Patient With Metabolic Syndrome
Brief Title: Vagal Nerve Stimulation as Therapeutic Approach on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rana Elbanna (Other)
Responsible Party: Sponsor-Investigator, Rana Elbanna, lecturer at faculty of physical therapy at Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003818
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus nerve stimulation group (Experimental): Vagus nerve stimulation group
  Interventions: Device: Vagal Stimulation; Other: Circuit training program
- Circuit weight training group Group (Experimental): Circuit weight training group Group
  Interventions: Other: Circuit training program

INTERVENTIONS:
Device: Vagal Stimulation — ear clips were placed in the ear region (auricular concha) at the stimulation site. The following stimulation settings were used: 1) density wave set to 20 Hz with a wave width of less than 1 ms; 2) intensity tuned to the patient's tolerance (4-6 mA)
  Arms: Vagus nerve stimulation group
Other: Circuit training program — The training regimen included ten different forms of resistance and aerobic exercise that were done three times a week for four weeks. The resistance training program included push-ups, squats, crunches, lunges, and a superman exercise program that included light jumping, jogging on the spot, foot stomping, steps, and jumping jacks

SUMMARY:
Participants were randomly assigned to two groups prior to their second visit: the Vagus nerve stimulation group (VNS) and the circuit training program. The randomization processes were conducted in Excel utilizing a random-number generator. Prior to the second visit, each participants' target exercise heart rate ranges were determined. Vagus nerve stimulation group(VNS) Patients rested on their sides in a sitting position. Following regular disinfection of the stimulation locations, ear clips were placed in the ear region (auricular concha) at the stimulation site. The training regimen included ten different forms of resistance and aerobic exercises.

DETAILED DESCRIPTION:
Vagus nerve stimulation group Group:

1. Each participant signed a consent form after receiving a detailed explanation about the procedure.
2. Patients rested on their sides in a sitting position.
3. Disinfection of the stimulation locations.
4. Ear clips were placed in the ear region (auricular concha) at the stimulation site.
5. Emotional eating was assessed by Emotional Eating Scale. 5. Patient satisfaction was assessed by The Short Assessment of Patient Satisfaction (SAPS).
6. Cortisol was assessed in lab. 7. After one month all the assessment procedure will be repeated again.

Circuit training group Group:

1. Each participant will signed a consent form after receiving a detailed explanation about the procedure.
2. The training regimen included ten different forms of resistance and aerobic exercises.
3. Emotional eating was assessed by Emotional Eating Scale.
4. Patient satisfaction was assessed by The Short Assessment of Patient Satisfaction (SAPS).

5 Cortisol was assessed in lab. 6. After one month all the assessment procedure will be repeated again.

ELIGIBILITY:
Inclusion Criteria:

having two or more than one of the following:

* Type 2 diabetes Miletus
* Hypertensive.
* Abnormal Cholesterol or Triglyceride level.
* BMI more than 30 kg/m
* Waist circumference more than 94 cm.

Exclusion Criteria:

* Vagotomy.
* Diathermy.
* Wallowing difficulties.
* Dyspnea.
* Cardiac arrhythmia.
* Seizure.
* Previous brain injury or surgery.
* Dysautonomia.

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Emotional eating | 4 weeks
  Emotional Eating was measured by a 15-item version of the Emotional Eating Scale. The scale required responses from 0 (no desire to eat) to 4 (an overwhelming urge to eat) based on "… the extent which the following feelings presently lead you to feel an urge to eat. A lower score indicated less of an urge to eat when the designated emotional state was present.
Patient satisfaction measures | 4 weeks
  The Short Assessment of Patient Satisfaction (SAPS) is a seven-item scale that can be utilized to measure patient satisfaction with their treatment.
  The seven-item Short Assessment of Patient Satisfaction (SAPS), which is scored on a 5-point scale (0-4) SAPS has a continuous score range of 0 to 28. SAPS categorical responses include 0-10 very dissatisfied, 11-18 dissatisfied, 19-26 satisfied, and 27-28 very satisfied.
Cortisol level | 4 weeks
  Participants use a disposable plastic straw to 'drool' saliva into the tube after collecting it in their mouths for a predetermined period of time (one minute) Saliva samples for cortisol measurement kept at room temperature until they are examined in a lab (4 to 6 hours)

SECONDARY OUTCOMES:
Body weight | 4 weeks
  After an eight-hour fast, body weight was taken between 7:00 and 10:00 am using a digital scale that was accurate to ±0.1 kg

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic faculty of physical therapy at Cairo University, Giza, Egypt

REFERENCES:
- [Derived] Elbanna RHM, Elabd SOA, Saleh MSM, Alghitany SIA. Effect of adding noninvasive auricular Vagal nerve stimulation to exercise program on emotional eating and stress responsiveness in patient with metabolic syndrome. Disabil Rehabil. 2025 Dec;47(24):6367-6374. doi: 10.1080/09638288.2025.2506824. Epub 2025 May 17. PMID 40382680